CLINICAL TRIAL: NCT03309566
Title: Bioequivalence Study of Efavirenz, Emtricitabine and Tenofovir in Healthy Volunteers, After Administering a Single Dose of a Fixed Dose Combination of the Test Formulation With Respect to the Reference Product, Atripla ® From Gador S.A
Brief Title: Bioequivalence Study of Two Formulatiosns With the Asscociaton of Efavirenz, Emtricitabine and Tenofovir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratorio Elea Phoenix S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRO-BEQ-EET-002-V.01
Record Dates: First submitted 2017-10-10; First posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Healthy
MeSH Terms: interventions — efavirenz; Tenofovir; Emtricitabine

STUDY DESIGN:
Intervention Model Description: Single-dose, two-way crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test - Reference (Experimental): A new formulation containing a combination of efavirenz 600 mg, emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg (T) followed by a branded formulation (R).
  Interventions: Drug: Efavirenz, tenofovir disoproxil fumarate and emtricitabine
- Reference - Test (Experimental): A branded formulation (R) followed by a new formulation containing a combination of efavirenz 600 mg, emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg (T).
  Interventions: Drug: Efavirenz, tenofovir disoproxil fumarate and emtricitabine

INTERVENTIONS:
Drug: Efavirenz, tenofovir disoproxil fumarate and emtricitabine — Two period administration of a formulation containing a combination of efavirenz 600 mg, emtricitabine 200 mg and tenofovir disoproxil fumarate 300 mg.

SUMMARY:
Bioequivalence study of two formulations containing a fixed dose combination of 600 mg Efavirenz, 200 mg Emtricitabine and 300 mg Tenofovir Disproxyl Fumarate in coated tablets under a single-dose, two-way crossover design.

ELIGIBILITY:
Inclusion Criteria:

Male subjects between 18 and 55 years. Subjects with body mass index (BMI) between 19 and 27 kg / m². Subjects whose complementary tests (ECG, blood and urine) are within normal and / or clinically insignificant according to the judgment of the investigator.

Subjects with systolic blood pressure between 110 mmHg and 139 mmHg; diastolic pressure between 70 mmHg and 89 mmHg; heart rate between 50 and 90 beats per minute.

Subjects who signed informed consent.

Exclusion Criteria:

Background of clinically significant allergies (except untreated asymptomatic seasonal allergies), drug hypersensitivity and / or hypersensitivity to any component of the formulations studied.

Drop of more than 20 mmHg in systolic blood pressure or more than 10 mmHg diastolic pressure in the first 3 minutes of postural change.

Active smoker more than 10 cigarettes / day. Pregnant or lactating women. Current clinical evidence of severe digestive disorders, surgery of the digestive tract (except appendectomy).

Current clinical evidence of kidney disease. Current evidence of liver disorders Current clinical evidence of respiratory and heart diseases. The presence of diabetes mellitus, thyroid dysfunction or other endocrine disorder.

Evidence of gastroduodenal disease. Current presence of any malignancy. History of abuse or addiction to drugs or alcohol during the past three years. Participation in a clinical trial within the last three months. Use of any drug within fourteen days before the start of the study. Subject donated or suffered blood loss during the last twelve weeks before the start of the study, or intends to donate blood within three months of the completion of the study.

Excessive drinking of tea, cocoa, mate, coffee and / or beverages containing caffeine (> 5 cups / day) or wine (> 0.5 L / day) or alcohol (> 50 ml / day).

ECG abnormalities. Positive serology for HIV, hepatitis B or hepatitis C.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-04 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-02-28 (Actual)

PRIMARY OUTCOMES:
Cmax | 192 hours
  Maximum plasma concentration
AUC | 192 hours
  Area under the curve

SECONDARY OUTCOMES:
Adverse events | 192 hours
  Drug related toxicity

CONTACTS AND LOCATIONS:
Overall Officials: María C Fritz, MD, Principal Investigator — DominguezLab
Locations (1):
- DominguezLab, Paraná, Entre Ríos Province, Argentina

IPD SHARING:
Plan to Share IPD: No